CLINICAL TRIAL: NCT07124598
Title: Virtual Intelligence for Transformative Lifestyle Solutions in Pain
Acronym: VITALS-Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); AugMend Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-16884; RM1DA055437 (NIH)
Record Dates: First submitted 2025-07-10; First posted 2025-08-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: Virtual Reality (VR)-based Chronic Pain Management; Opioid Management; Opioid Use Disorder; Artificial Intelligence (AI)
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study represents exploratory research comparing assessment methodologies rather than clinical implementation of a diagnostic tool. The breadth of comparison domains and focus on methodology validation supports the research-oriented, non-diagnostic nature of the application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-guided Virtual Reality (VR) Session (Experimental): The intervention is a single-day 45-minute VR intervention which is subdivided into 3 smaller sessions:
  Session 1: A 15-minute AI check-in to ask questions about biopsychosocial health Session 2: A 20-minute Pain Coping Skills Training (PCST) session offering psychoeducation on managing chronic pain Session 3: A 10-minute stress reduction exercise.
  Interventions: Device: VR Headset Device - Meta Quest 3

INTERVENTIONS:
Device: VR Headset Device - Meta Quest 3 — The VR sessions will be conducted using hardware and software developed by AugMend Health Company. The AI-guided sessions will be administered using the commercially available Meta Quest 3 headset, which delivers high-resolution VR images and spatial audio through a standalone, wireless system.

SUMMARY:
This pilot study aims to evaluate the feasibility and acceptability of a VR-based chronic pain management intervention with a virtual AI coach for patients with Opioid misuse and opioid use disorder (OM/OUD). The intervention is a single-day 45-minute VR intervention which is subdivided into three smaller sessions:

Session 1: A 15-minute AI check-in to ask questions about biopsychosocial health, Session 2: A 20-minute Pain Coping Skills Training (PCST) session offering psychoeducation on managing chronic pain Session 3: A 10-minute stress reduction exercise.

The VR sessions will be conducted using hardware (VR Headset Device - Meta Quest 3) and software developed by AugMend Health Company.

The study will be conducted in a clinical setting at the Montefiore Multidisciplinary Pain Medicine Program (MMPP), a Pain Medicine outpatient specialty practice within a major urban medical center. MMPP providers see thousands of patients every month, some of which have concurrent opioid misuse or OM/OUD.

DETAILED DESCRIPTION:
Opioid misuse and opioid use disorder (OM/OUD) constitute a persistent public health emergency that is projected to escalate. In 2018, about 2 million individuals in the US had an OM/OUD, associated with a high mortality rate of approximately 130 daily deaths, comorbid psychiatric disorders, and other poor health outcomes. Further interventions are needed to reduce the impact of opioid misuse, OM/OUD, and overdose. Chronic pain affects over 100 million individuals in the United States, and opioids prescribed to treat pain can increase risks of misuse, physiological dependence, and OM/OUD. Research indicates that 64.4% of OM/OUD patients report chronic pain, which can trigger relapse, reduce adherence to OM/OUD treatment, and diminish quality of life. Standard care for OM/OUD includes medication, such as methadone maintenance therapy (MMT), and psychosocial treatment. Given the adverse effects of chronic pain among patients with OM/OUD, there is an unmet need for complementary approaches to assist OM/OUD patients with pain.

In patients with OM/OUD and Chronic pain, psychosocial treatment is provided using a variety of approaches, one of which is Cognitive behavioral therapy (CBT). CBT is an evidence-based treatment that has been shown to be effective in managing both chronic pain and OM/OUD by helping patients develop coping strategies and alter maladaptive thought patterns. However, traditional CBT faces challenges such as limited accessibility due to geographic, socioeconomic, and psychological barriers, and high dropout rates due to its repetitive nature. Studies show patient-reported barriers to use of non-pharmacological treatments in chronic pain included high cost, transportation problems and low motivation, while top-ranked facilitators included availability of a wider array of options and a team-based approach that included follow-up. For this reason, more readily available and accessible options are needed.

VR technology offers an innovative treatment paradigm for patients with OM/OUD and chronic pain. A recent study showed that a VR meditative intervention can modulate pain and modify neurobiological markers in patients with OM/OUD. The immersive environment can significantly enhance patient engagement, making sessions more interactive and enjoyable, while providing pain relief. Furthermore, by providing a captivating virtual experience, VR-based psychosocial check ins can improve retention rates and ensure patients complete their therapeutic programs.

A significant innovation of VR-based biopsychosocial check-ins is its potential to make psychosocial interventions more accessible and tailored to individual needs. Traditional face-to-face CBT can be inaccessible due to geographic, socioeconomic, and psychological barriers. VR can overcome these barriers by providing a flexible treatment option within the clinical setting. Moreover, VR environments can be customized to accommodate patients with varying literacy levels, using visual aids and interactive elements to ensure comprehension and engagement, particularly for those with a third-grade reading level. VR provides an experiential learning platform where patients can practice biopsychosocial skills in a controlled, simulated environment. This method allows for repeated practice of coping strategies and pain management techniques, which is crucial for skill acquisition and generalization to real-world settings. The ability to engage in realistic scenarios within VR can enhance the transfer of these skills to daily life, improving patients' ability to manage pain and opioid cravings outside the clinical setting.

Few studies have previously utilized VR and AI to deliver conversational biopsychosocial check ins and lifestyle education specifically targeting the combined treatment of chronic pain and OM/OUD. There are limited studies on the efficacy of AI tools in mental health. Mental Health America has an AI-powered tool which allows users to type their negative thoughts, and the program assists them in reframing the thoughts. This novel application not only addresses the limitations of traditional CBT but also explores the potential of VR and AI as a versatile and effective medium for treating co-occurring conditions. The integration of VR and AI represents a promising approach that could significantly enhance therapeutic outcomes for patients with these complex conditions. The AI virtual coach is designed to provide a non-judgmental, empathetic, and supportive environment. By interacting with an AI coach, patients may feel more comfortable discussing sensitive issues without fear of judgment or bias, which can reduce internalized stigma and encourage openness. Additionally, some patients find it easier to disclose information to AI-based avatars. AI systems can enhance patient support by providing adaptive treatment recommendations based on patient feedback, effectively supporting patients and optimizing healthcare resources. Moreover, AI allows the adaptivity of the difficulty level to the demographic specificity of the patient, ensuring a more personalized and effective treatment approach. Research has shown that interactive and immersive environments can significantly enhance user engagement, leading to better adherence to treatment protocols. To promote equitable access to our VR intervention, the investigator team anticipates expanding its availability for in-home use in future phases and larger studies as part of the research. By developing portable and user-friendly VR systems, the study team aims to overcome barriers such as transportation difficulties and limited access to clinical facilities, particularly for underserved populations. This approach aligns with research indicating that home-based VR interventions can effectively reach diverse patient populations and improve accessibility to care.

The VR software has been determined to be non-significant risk by the Institutional Review Board (IRB) based on the 21st Century Cures Act. Section 520(o)(1) of the Food Drug and Cosmetic (FD&C) Act specifically excludes certain software functions from medical device classification.

ELIGIBILITY:
Inclusion Criteria:

* Patients with opioid misuse or International Classification of Diseases 10th revision (ICD-10) diagnosis of opioid use disorder
* Patients with Chronic pain of at least moderate intensity (>4 Pain Intensity Score) with no pain medication changes in 14 days
* Ability to understand written/spoken instruction and provide informed consent in English
* Ability and willingness to participate in all components of the study

Exclusion Criteria:

* History of severe motion sickness, cybersickness, or conditions that could make participation in VR hazardous or cause adverse effects
* Conditions that could prevent proper use of VR headset (such as vision problems that cannot be corrected by contact lenses or glasses that fit in VR, Significant hearing impairments that cannot be corrected by a hearing device)
* History of seizures or seizure disorder
* Acute exacerbation of psychiatric conditions that preclude the ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment Rate | Approximately 6 months
  Feasibility of the intervention will be assessed by tracking and determining the recruitment rate for the study. For purposes of this study recruitment rate will be defined as the number/percentage of participants who are consented, screened, and enrolled over the 6-month timeframe will be summarized and reported.
Feasibility - Completion | Approximately 6 months
  Feasibility of the intervention will also be assessed by the number/percentage of participants who are able to successfully complete all three AI-guided, VR sessions. The number/percentage of participants that complete all three sessions will be summarized and reported using basic descriptive statistics.
Feasibility - Virtual Reality Experience and Feasibility Survey (VREFS) | Up to 1 hour following completion of ~ 45-minute VR session
  Feasibility of the intervention as assessed by VREFS will also be determined. The VREFS is a comprehensive feasibility tool which measures feasibility across 7 distinct dimensions: Core Therapeutic Alliance (6 items); Cultural Competence & Identity (5 items); Continuity & Future Use (3 items); Privacy & Trust (8 items); Medical Trust (3 items); Usability (11 items); and Overall Experience (6 items). The survey also consists of 4 additional items and 6 avatar-specific items. Participants are asked to evaluate and rate each statement on a 7-point scale ranging from 1 ("Strongly disagree") to 7 ("Strongly agree") such that higher scores are associated with a more favorable assessment of the intervention and study. Results will be summarized and reported using basic descriptive statistics.
Acceptability - Acceptability of Intervention Measure (AIM) | Up to 1 hour following completion of ~ 45-minute VR session
  Acceptability of the intervention will be evaluated using AIM. AIM consists of 4 statements which asks participants to rate the acceptability of the intervention measures on a 5-point scale ranging from 1 ("Completely disagree") to 5 ("Completely agree") for an overall possible scoring range of 4-20, with higher scores being indicative of greater acceptability of the measures. Results will be summarized using basic descriptive statistics.
Satisfaction - Change | Up to 1 hour following completion of ~ 45-minute VR session
  Satisfaction will be measured and assessed using the Patient's Global Impression of Change Scale (PGIC) questionnaire completed following the VR intervention. Participants will be asked to respond to the following query, "Since beginning treatment at this clinic, how would you describe the change (if any) in Activity, Limitations, Symptoms, Emotions and Overall Quality of Life, related to your painful condition? (tick only 1 box)" on a 7-point Likert scale ranging from 1 - "No change (or condition is worse)" to 7 "A great deal better, and a considerable improvement that has made all the difference" such that higher scores are associated with improved global impression of change. Results will be summarized using basic descriptive statistics.
Satisfaction - Degree of Change | Up to 1 hour following completion of ~ 45-minute VR session
  Satisfaction will be also measured and assessed using the following question derived from the PGIC questionnaire: "In a similar way, please circle the number below that matches your degree of change since beginning care at this clinic." Participants will be asked to rate the degree of change on an 11-point scale ranging from 0 ("Much better") to 10 ("Much worse") such that lower scores are associated with a worsened degree of change. Results will be summarized using basic descriptive statistics.

SECONDARY OUTCOMES:
Efficacy - Change in Pain Severity Level | From pre- to post-VR session, up to 4 hours
  Change in pain severity will be assessed based on the Visual Analog Scale (VAS) administered prior to and following the VR session. Participants will be asked to rate their average pain over the last 24 hours below by selecting a number that describes their pain level on an 11-point Likert scale ranging from 0 ("NO pain") to 10 (WORST imaginable pain"). Higher VAS scores are associated with greater pain intensity/severity. For purposes of this study change in pain severity from pre- to post-VR session will be assessed and negative scores will be associated with decreased pain severity from pre- to post-intervention. Results will be summarized using basic descriptive statistics and analyzed by paired t-tests or Wilcoxon signed-rank tests.
Efficacy - Change in Anxiety Level | From pre- to post-VR session, up to 4 hours
  Change in anxiety will be assessed using the Pain Anxiety Symptom Scale Short Form 20 (PASS-20) administered prior to and following the VR session. The PASS-20 is a 20-item questionnaire that assesses pain-related anxiety. Participants will be asked to rate each of the 20 items on the questionnaire in terms of frequency on a 6-point Likert scale ranging from 0 ("Never") to 5 ("Always"). Higher PASS-20 scores are associated with greater pain-related anxiety. For purposes of this study change in anxiety from pre- to post-VR session will be assessed and negative scores will be associated with decreased pain-related anxiety from pre- to post-intervention. Results will be summarized using basic descriptive statistics and analyzed by paired t-tests or Wilcoxon signed-rank tests.
Efficacy - Self-efficacy in managing Drug/Opioid use and cravings | From pre- to post-VR session, up to 4 hours
  Self-efficacy in managing Drug/Opioid use and cravings will be evaluated using the Drug Abstinence Self-Efficacy Scale (DASES) administered prior to and following the VR session. DASES describes 16 situations that may trigger someone's intention to take drugs and asks participants to select a response indicating what they would be likely to do in each situation. Participants are asked to rate each of the 16 situations using a 7-point scale ranging from 1 ("Certainly no") to 7 ("Certainly yes") such that higher scores are indicative of an individual having more confidence in their ability to resist drug use in specific situations. For purposes of this study change in self-efficacy from pre- to post-VR session will be assessed and positive scores will be associated with increased self-efficacy from pre- to post-intervention. Results will be summarized using basic descriptive statistics and analyzed by paired t-tests or Wilcoxon signed-rank tests.
Safety - Virtual Reality Sickness Questionnaire (VRSQ) | Up to 1 hour following completion of ~ 45-minute VR session
  Safety will be assessed using the VRSQ. The VRSQ outlines 9 symptoms (General discomfort, Fatigue, Headache, Eye strain, Difficulty focusing, Fullness of the Head, Blurred vision, Dizziness with eyes closed, and Vertigo) and asks participants to rate how much each symptom is affecting them at the time of the study as follows: 0 = None, 1 = Slight, 2 = Moderate, 3 = Severe. Scoring is determined by summing the score of the first four symptoms on the list (=A); summing the score of the last 5 symptoms on the list (=B); calculating the variable "C" in C = A/12 x 100; and calculating the variable "D" in D = B/15 x100. Finally, A VRSQ score is determined by the following formula: VRSQ = (C+D)/2. Higher VRSQ scores are indicative of greater levels of VR sickness. Results will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Moorice A Caparo, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Multidisciplinary Pain Medicine Program (MMPP) at Montefiore Einstein Hutchinson Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scholl L, Seth P, Kariisa M, Wilson N, Baldwin G. Drug and Opioid-Involved Overdose Deaths - United States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2018 Jan 4;67(5152):1419-1427. doi: 10.15585/mmwr.mm675152e1. PMID 30605448
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] Florence CS, Zhou C, Luo F, Xu L. The Economic Burden of Prescription Opioid Overdose, Abuse, and Dependence in the United States, 2013. Med Care. 2016 Oct;54(10):901-6. doi: 10.1097/MLR.0000000000000625. PMID 27623005
- [Background] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Background] Ehde DM, Dillworth TM, Turner JA. Cognitive-behavioral therapy for individuals with chronic pain: efficacy, innovations, and directions for research. Am Psychol. 2014 Feb-Mar;69(2):153-66. doi: 10.1037/a0035747. PMID 24547801
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Freeman D, Reeve S, Robinson A, Ehlers A, Clark D, Spanlang B, Slater M. Virtual reality in the assessment, understanding, and treatment of mental health disorders. Psychol Med. 2017 Oct;47(14):2393-2400. doi: 10.1017/S003329171700040X. Epub 2017 Mar 22. PMID 28325167
- [Background] Garcia AN, Kelley ML, Rentz TO, Lee SS, Donaldson D, Borrego J. Feasibility of a virtual reality intervention for the treatment of pediatric pain and anxiety during burn wound care. J Burn Care Res. 2022;43(1):46-55.
- [Background] Dutra L, Stathopoulou G, Basden SL, Leyro TM, Powers MB, Otto MW. A meta-analytic review of psychosocial interventions for substance use disorders. Am J Psychiatry. 2008 Feb;165(2):179-87. doi: 10.1176/appi.ajp.2007.06111851. Epub 2008 Jan 15. PMID 18198270
- [Background] Andersson G, Cuijpers P, Carlbring P, Riper H, Hedman E. Guided Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: a systematic review and meta-analysis. World Psychiatry. 2014 Oct;13(3):288-95. doi: 10.1002/wps.20151. PMID 25273302
- [Background] Bouchard S, Renaud P, Cournoyer LG. Revising the usability of a virtual reality cognitive-behavioral therapy for subthreshold autism. Cyberpsychol Behav Soc Netw. 2012;15(8):481-488.
- [Background] Becker WC, Dorflinger L, Edmond SN, Islam L, Heapy AA, Fraenkel L. Barriers and facilitators to use of non-pharmacological treatments in chronic pain. BMC Fam Pract. 2017 Mar 20;18(1):41. doi: 10.1186/s12875-017-0608-2. PMID 28320337
- [Background] Segawa T, Baudry T, Bourla A, Blanc JV, Peretti CS, Mouchabac S, Ferreri F. Virtual Reality (VR) in Assessment and Treatment of Addictive Disorders: A Systematic Review. Front Neurosci. 2020 Jan 10;13:1409. doi: 10.3389/fnins.2019.01409. eCollection 2019. PMID 31998066
- [Background] Garcia-Palacios A, Botella C, Hoffman H, Fabregat S. Comparing acceptance and refusal rates of virtual reality exposure vs. in vivo exposure by patients with specific phobias. Cyberpsychol Behav. 2007 Oct;10(5):722-4. doi: 10.1089/cpb.2007.9962. PMID 17927544
- [Background] Gerardi M, Cukor J, Difede J, Rizzo A, Rothbaum BO. Virtual reality exposure therapy for post-traumatic stress disorder and other anxiety disorders. Curr Psychiatry Rep. 2010 Aug;12(4):298-305. doi: 10.1007/s11920-010-0128-4. PMID 20535592
- [Background] Triberti S, Repetto C, Riva G. Psychological factors influencing the effectiveness of virtual reality-based analgesia: a systematic review. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):335-45. doi: 10.1089/cyber.2014.0054. PMID 24892195
- [Background] Austin PD, Siddall PJ. Virtual reality for the treatment of neuropathic pain in people with spinal cord injuries: A scoping review. J Spinal Cord Med. 2021 Jan;44(1):8-18. doi: 10.1080/10790268.2019.1575554. Epub 2019 Feb 1. PMID 30707649
- [Background] Austin PD, Siddall PJ, Lovell MR. Feasibility and acceptability of virtual reality for cancer pain in people receiving palliative care: a randomised cross-over study. Support Care Cancer. 2022 May;30(5):3995-4005. doi: 10.1007/s00520-022-06824-x. Epub 2022 Jan 21. PMID 35064330
- [Background] Cukor J, Spitalnick J, Difede J, Rizzo A, Rothbaum BO. Emerging treatments for PTSD. Clin Psychol Rev. 2009 Dec;29(8):715-26. doi: 10.1016/j.cpr.2009.09.001. Epub 2009 Sep 10. PMID 19800725
- [Background] Newman MG, Szkodny LE, Llera SJ, Przeworski A. A review of technology-assisted self-help and minimal contact therapies for anxiety and depression: is human contact necessary for therapeutic efficacy? Clin Psychol Rev. 2011 Feb;31(1):89-103. doi: 10.1016/j.cpr.2010.09.008. Epub 2010 Oct 14. PMID 21130939
- [Background] Wiederhold BK, Wiederhold MD. Virtual reality for posttraumatic stress disorder and stress inoculation training. J Cyber Ther Rehabil. 2005;2(4):117-127.
- [Background] Rothbaum BO, Hodges L, Smith S, Lee JH, Price L. A controlled study of virtual reality exposure therapy for the fear of flying. J Consult Clin Psychol. 2000 Dec;68(6):1020-6. doi: 10.1037//0022-006x.68.6.1020. PMID 11142535
- [Background] Morina N, Ijntema H, Meyerbroker K, Emmelkamp PM. Can virtual reality exposure therapy gains be generalized to real-life? A meta-analysis of studies applying behavioral assessments. Behav Res Ther. 2015 Nov;74:18-24. doi: 10.1016/j.brat.2015.08.010. Epub 2015 Aug 31. PMID 26355646
- [Background] Levin ME, Hayes SC, Pistorello J, Seeley JR. Web-Based Self-Help for Preventing Mental Health Problems in Universities: Comparing Acceptance and Commitment Training to Mental Health Education. J Clin Psychol. 2016 Mar;72(3):207-25. doi: 10.1002/jclp.22254. Epub 2016 Jan 19. PMID 26784010
- [Background] Changing Thoughts with an AI Assistant. Mental Health America. https://screening.mhanational.org/changing-thoughts-with-an-ai-assistant/
- [Background] Maddox T, Garcia H, Ffrench K, Maddox R, Garcia L, Krishnamurthy P, Okhotin D, Sparks C, Oldstone L, Birckhead B, Sackman J, Mackey I, Louis R, Salmasi V, Oyao A, Darnall BD. In-home virtual reality program for chronic low back pain: durability of a randomized, placebo-controlled clinical trial to 18 months post-treatment. Reg Anesth Pain Med. 2024 May 7;49(5):373-375. doi: 10.1136/rapm-2022-104093. No abstract available. PMID 36427904
- [Background] Lucas, Gale M., et al. "It's Only a Computer: Virtual Humans Increase Willingness to Disclose." Computers in Human Behavior, vol. 37, Aug. 2014, pp. 94-100, https://doi.org/10.1016/j.chb.2014.04.043.
- [Background] Rogers, Shane L., et al. "Realistic Motion Avatars Are the Future for Social Interaction in Virtual Reality." Frontiers in Virtual Reality, vol. 2, 3 Jan. 2022, https://doi.org/10.3389/frvir.2021.750729.
- [Background] Pauw, Lisanne S., et al. "The Avatar Will See You Now: Support from a Virtual Human Provides Socio-Emotional Benefits." Computers in Human Behavior, vol. 136, Nov. 2022, p. 107368, https://doi.org/10.1016/j.chb.2022.107368.